CLINICAL TRIAL: NCT02823574
Title: A Double-Blind, Randomized, Two Arm Phase 2 Study of Nivolumab in Combination With Ipilimumab Versus Nivolumab in Combination With Ipilimumab Placebo in Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Study of Nivolumab in Combination With Ipilimumab Versus Nivolumab in Combination With Ipilimumab Placebo in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Acronym: CheckMate 714
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA209-714; 2016-001645-64 (EudraCT Number)
Expanded Access: NCT03126643 (Approved for marketing)
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Results first posted 2022-04-21 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab and Ipilimumab (Experimental): Specified dose on specified days
  Interventions: Biological: Nivolumab; Biological: Ipilimumab
- Nivolumab and Ipilimumab-placebo (Active Comparator): Specified dose on specified days
  Interventions: Biological: Nivolumab; Other: Placebo

INTERVENTIONS:
Biological: Nivolumab
  Other Names: Opdivo
Biological: Ipilimumab
  Arms: Nivolumab and Ipilimumab
Other: Placebo
  Arms: Nivolumab and Ipilimumab-placebo

SUMMARY:
A study in patients with metastatic or recurrent squamous cell cancer of the head and neck to evaluate the effectiveness of Nivolumab plus Ipilumumab vs. Nivolumab alone (CheckMate 714)

ELIGIBILITY:
Inclusion Criteria:

* Confirmed squamous cell head and neck cancer
* Widespread (metastatic) disease, or returned after previous treatment (recurrent)
* Tumor sample must be available for analysis of PDL1 (Programmed death-ligand 1) and HPV [Human Papilloma Virus (oropharynx only)]
* Performance status ECOG 0-1 (Eastern Cooperative Oncology Group)

Exclusion Criteria:

* Previous treatment for metastatic or recurrent disease
* Cancer arising from one of the following primary sites: paranasal sinus, nasopharynx, salivary gland, skin
* Any non-squamous subtype
* Active autoimmune disease
* Positive test for hepatitis B, C or HIV (Human Immunodeficiency Virus) virus
* Previous treatment with checkpoint inhibitor drugs
* Active CNS metastases or carcinomatous meningitis

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2016-11-08 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (105):
- United States (28):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Local Institution - 0034, Duarte, California
  - Los Angeles Cancer Network, Los Angeles, California
  - Ucla Department Of Medicine, Los Angeles, California
  - Local Institution - 0098, Redondo Beach, California
  - Local Institution - 0004, Sacramento, California
  - Local Institution - 0072, San Francisco, California
  - Local Institution - 0097, San Luis Obispo, California
  - Central Coast Med Oncology, Santa Maria, California
  - Local Institution - 0101, New Haven, Connecticut
  - Local Institution - 0007, Tampa, Florida
  - Local Institution - 0010, Atlanta, Georgia
  - Local Institution - 0015, Decatur, Georgia
  - Local Institution - 0087, Chicago, Illinois
  - Ft. Wayne Med Onco-Hema Inc, Fort Wayne, Indiana
  - Local Institution - 0005, Louisville, Kentucky
  - Oncology Associated Of Western Kentucky, Paducah, Kentucky
  - Local Institution - 0001, Boston, Massachusetts
  - Local Institution - 0071, Boston, Massachusetts
  - Local Institution - 0042, Rochester, Minnesota
  - Mission Hospital, Inc, Asheville, North Carolina
  - Local Institution - 0103, Cincinnati, Ohio
  - Local Institution - 0070, Cleveland, Ohio
  - Local Institution - 0008, Portland, Oregon
  - Local Institution - 0006, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation, Sayre, Pennsylvania
  - Local Institution - 0102, Dallas, Texas
  - Local Institution - 0038, Seattle, Washington
- Argentina (2):
  - Local Institution - 0121, Pergamino, Buenos Aires
  - Local Institution - 0111, Buenos Aires
- Belgium (3):
  - Local Institution - 0023, Ghent
  - Local Institution - 0074, Sint-Niklaas
  - Local Institution - 0053, Yvoir
- Brazil (12):
  - Local Institution - 0046, Belo Horizonte, Minas Gerais
  - Local Institution - 0124, Ipatinga, Minas Gerais
  - Local Institution - 0047, Curitiba, Paraná
  - Local Institution - 0125, Caxias do Sul, Rio Grande do Sul
  - Local Institution - 0051, Ijuí, Rio Grande do Sul
  - Local Institution - 0052, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0045, Barretos, São Paulo
  - Local Institution - 0123, Santo André, São Paulo
  - Local Institution - 0048, São José do Rio Preto, São Paulo
  - Local Institution, Rio de Janeiro
  - Local Institution - 0049, São Paulo
  - Local Institution - 0050, São Paulo
- Canada (5):
  - Local Institution - 0013, Edmonton, Alberta
  - Local Institution - 0056, Ottawa, Ontario
  - Local Institution - 0012, Toronto, Ontario
  - Local Institution - 0016, Montreal, Quebec
  - Local Institution - 0014, Québec, Quebec
- Local Institution - 0115, Santiago, Santiago Metropolitan, Chile
- Czechia (3):
  - Local Institution - 0022, Brno
  - Local Institution - 0020, Hradec Králové
  - Local Institution - 0021, Olomouc
- Local Institution - 0069, Helsinki, Finland
- France (9):
  - Local Institution - 0032, Amiens
  - Local Institution - 0120, Bordeaux
  - Local Institution - 0073, Clermont-Ferrand
  - Local Institution - 0089, Clichy
  - Local Institution - 0029, Lyon
  - Local Institution - 0075, Marseille
  - Local Institution - 0079, Nice
  - Local Institution - 0030, Rennes
  - Local Institution - 0088, Villejuif
- Local Institution - 0026, Dublin, Dublin, Ireland
- Italy (2):
  - Local Institution, Milan
  - Local Institution - 0119, Napoli
- Mexico (3):
  - Local Institution - 0090, Mérida, Yucatán
  - Local Institution - 0107, Mérida, Yucatán
  - Local Institution - 0108, Oaxaca City
- Netherlands (3):
  - Local Institution - 0068, Amsterdam
  - Local Institution - 0028, Amsterdam
  - Local Institution - 0027, Groningen
- Norway (2):
  - Local Institution - 0065, Bergen
  - Local Institution - 0064, Oslo
- Romania (5):
  - Local Institution - 0055, Bucharest
  - Local Institution - 0054, Cluj-Napoca
  - Local Institution - 0033, Craiova
  - Local Institution - 0060, Iași
  - Local Institution - 0059, Suceava
- Russia (2):
  - Local Institution - 0031, Moscow
  - Local Institution - 0092, Ryazan
- South Africa (4):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Pretoria, Gauteng
  - Local Institution - 0017, Sandton, Gauteng
  - Local Institution, Cape Town, Western Cape
- Spain (6):
  - Local Institution - 0040, A Coruña
  - Local Institution - 0116, Barcelona
  - Local Institution - 0039, Barcelona
  - Local Institution - 0077, Madrid
  - Local Institution - 0076, Marbella
  - Local Institution - 0041, San Sabastian Gipuzkoa
- Sweden (3):
  - Local Institution - 0067, Gothenburg
  - Local Institution - 0037, Lund
  - Local Institution - 0035, Stockholm
- Turkey (Türkiye) (3):
  - Local Institution - 0063, Adana
  - Local Institution - 0066, Antalya
  - Local Institution - 0062, Izmir
- United Kingdom (7):
  - Local Institution - 0110, Aberdeen, Aberdeenshire
  - Local Institution - 0086, London, Greater London
  - Local Institution - 0083, Metropolitan Borough of Wirral, Merseyside
  - Local Institution - 0081, Sutton, Surrey
  - Local Institution - 0114, Cardiff
  - Local Institution - 0084, Glasgow
  - Local Institution - 0082, Newcastle upon Tyne

REFERENCES:
- [Derived] Harrington KJ, Ferris RL, Gillison M, Tahara M, Argiris A, Fayette J, Schenker M, Bratland A, Walker JWT, Grell P, Even C, Chung CH, Redman R, Coutte A, Salas S, Grant C, de Azevedo S, Soulieres D, Hansen AR, Wei L, Khan TA, Miller-Moslin K, Roberts M, Haddad R. Efficacy and Safety of Nivolumab Plus Ipilimumab vs Nivolumab Alone for Treatment of Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck: The Phase 2 CheckMate 714 Randomized Clinical Trial. JAMA Oncol. 2023 Jun 1;9(6):779-789. doi: 10.1001/jamaoncol.2023.0147. PMID 37022706
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 425 randomized and 423 participants treated.
Groups:
- Treatment A - Platinum Refractory Subgroup: Participants with histologically confirmed Squamous Cell Carcinoma of the Head and Neck (SCCHN) that has recurred during or less than 6 months after completion of previous platinum-based chemotherapy.
  Treated with Nivolumab 3 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W
- Treatment B - Platinum Refractory Subgroup: Participants with histologically confirmed Squamous Cell Carcinoma of the Head and Neck (SCCHN) that has recurred during or less than 6 months after completion of previous platinum-based chemotherapy.
  Treated with Nivolumab 3 mg/kg Q2W + Ipilimumab-Placebo Q6W
- Treatment A - Platinum Eligible Subgroup: Participants with histologically confirmed Squamous Cell Carcinoma of the Head and Neck (SCCHN) who are platinum naive or have recurred 6 months or more after completion of previous platinum-based chemotherapy.
  Treated with Nivolumab 3 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W
- Treatment B - Platinum Eligible Subgroup: Participants with histologically confirmed Squamous Cell Carcinoma of the Head and Neck (SCCHN) who are platinum naive or have recurred 6 months or more after completion of previous platinum-based chemotherapy.
  Treated with Nivolumab 3 mg/kg Q2W + Ipilimumab-Placebo Q6W
Period: Randomization
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Started | 159 | 82 | 123 | 61
Completed (Continuing to Treatment Period) | 158 | 82 | 122 | 61
Not Completed | 1 | 0 | 1 | 0
Not completed — Disease Progression | 0 | 0 | 1 | 0
Not completed — AE unrelated to Study Drug | 1 | 0 | 0 | 0
Period: Treatment Period
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Started | 158 | 82 | 122 | 61
Completed (Completed = Continuing in the Treatment Period) | 0 | 0 | 0 | 0
Not Completed | 158 | 82 | 122 | 61
Not completed — Poor/Non Compliance | 1 | 0 | 0 | 1
Not completed — Maximum Clinical Benefit | 8 | 4 | 7 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Participant withdrew consent | 4 | 0 | 0 | 1
Not completed — Participant request to discontinue | 5 | 0 | 3 | 2
Not completed — Adverse Event unrelated to to study Drug | 10 | 2 | 9 | 2
Not completed — Study Drug Toxicity | 11 | 2 | 14 | 4
Not completed — Disease Progression | 113 | 64 | 82 | 43
Not completed — Other reasons | 5 | 9 | 3 | 6
Not completed — Participant no longer meets study criteria | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup | Total
Number analyzed (Participants) | 159 | 82 | 123 | 61 | 425
Age, Categorical [Count of Participants; unit: Participants] — Population: All Randomized Participants is the total of the 2 subgroups
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 119 | 63 | 79 | 40 | 301
    >=65 years | 40 | 19 | 44 | 21 | 124
Sex: Female, Male [Count of Participants; unit: Participants] — Population: All Randomized Participants is the total of the 2 subgroups
  Participants
    Female | 29 | 18 | 18 | 14 | 79
    Male | 130 | 64 | 105 | 47 | 346
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Randomized Participants is the total of the 2 subgroups
  Participants
    Hispanic or Latino | 10 | 7 | 6 | 6 | 29
    Not Hispanic or Latino | 56 | 23 | 66 | 25 | 170
    Unknown or Not Reported | 93 | 52 | 51 | 30 | 226
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: All Randomized Participants is the total of the 2 subgroups
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 3 | 1 | 0 | 1 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 2 | 3 | 2 | 1 | 8
    White | 141 | 75 | 120 | 58 | 394
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 13 | 3 | 1 | 1 | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Refractory Subgroup
Description: ORR is defined as best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized participants for each treatment group.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Approximately up to 30 months (from FPFV to Data base lock)
Population: All Randomized Participants - Platinum Refractory Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
percentage of participants | 13.2 [8.4 to 19.5] | 18.3 [10.6 to 28.4]
Statistical Analysis 1: Comparison: Treatment A - Platinum Refractory Subgroup vs Treatment B - Platinum Refractory Subgroup; Treatment A over Treatment B; Test type: Superiority; p = 0.2897, Mantel Haenszel; Odds Ratio (OR) = 0.68, 95.5% CI 2-sided [0.33 to 1.43]

2. Primary Outcome: Duration of Response (DOR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Refractory Subgroup
Description: The time between the date of first confirmed response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first.
Time Frame: Approximately up to 30 months (from FPFV to Data base lock)
Population: Platinum Refractory Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 21 | 15
Months | NA [11.01 to NA] — Insufficient number of events for median, upper limit not calculable | 11.07 [4.14 to NA] — upper limit not calculable

3. Primary Outcome: Time to Response (TTR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Refractory Subgroup
Description: Time to Response (TTR) for participants demonstrating a response (either CR or PR) was defined as the time from the date of randomization to the date of the first confirmed response.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Approximately up to 30 months (from FPFV to Data base lock)
Population: Platinum refractory responders
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 21 | 15
Months | 2.56 [1.1 to 6.6] | 1.51 [1.2 to 7.7]

4. Secondary Outcome: Objective Response Rate (ORR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Eligible Subgroup
Description: ORR is defined as percentage of participants with a complete response (CR) or partial response (PR).
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to end of study. Approximately 63 Months
Population: All Randomized Participants - Platinum Eligible Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
percentage of participants | 20.3 [13.6 to 28.5] | 29.5 [18.5 to 42.6]

5. Secondary Outcome: Duration of Response (DOR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Eligible Subgroup
Description: as for outcome 2
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum eligible subgroup responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 25 | 18
Months | 27.04 [11.01 to NA] — Insufficient number of events for median, upper limit not calculable | 24.61 [6.90 to NA] — Insufficient number of events for median, upper limit not calculable

6. Secondary Outcome: Progression Free Survival (PFS) as Determined by Blinded Independent Central Review (BIRC) - Platinum Refractory Subgroup
Description: The time from randomization to the date of first documented disease progression, or death due to any cause, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum Refractory subgroup all randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months | 2.50 [1.45 to 2.76] | 2.60 [1.54 to 3.38]
Statistical Analysis 1: Comparison: Treatment A - Platinum Refractory Subgroup vs Treatment B - Platinum Refractory Subgroup; Test type: Superiority; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.78 to 1.41] — computed using a cox proportional hazard model stratified by randomization PD-L1 and HPV status

7. Secondary Outcome: Progression Free Survival (PFS) as Determined by Blinded Independent Central Review (BIRC) - Platinum Eligible Subgroup
Description: as for outcome 6
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum Eligible subgroup all randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
Months | 2.76 [1.64 to 4.17] | 2.86 [1.51 to 5.65]
Statistical Analysis 1: Comparison: Treatment A - Platinum Eligible Subgroup vs Treatment B - Platinum Eligible Subgroup; Test type: Superiority; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.78 to 1.41] — computed using a cox proportional hazard model stratified by randomization PDL-1 and HPV status

8. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to the date of death from any cause. Participants were censored at the date they were last known to be alive and at the date of randomization if they were randomized but had no follow-up.
Time Frame: From randomization to death. Approximately 63 Months
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment A: Participants in both Platinum Refractory Subgroup and Platinum Eligible Subgroup treated with Nivolumab 3 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W
- Treatment B: Participants in both Platinum Refractory Subgroup and Platinum Eligible Subgroup treated with Nivolumab 3 mg/kg Q2W + Ipilimumab-Placebo Q6W
Arm/Group | Treatment A | Treatment B
Number analyzed (Participants) | 282 | 143
Months | 9.76 [7.52 to 11.47] | 11.30 [8.48 to 14.00]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Superiority; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.87 to 1.36] — computed using a cox proportional hazard model stratified by randomization PDL-1 and HPV status

9. Secondary Outcome: Overall Survival (OS) - Platinum Refractory Subgroup
Description: as for outcome 8
Time Frame: From randomization to death. Approximately 63 Months
Population: All Randomized Participants - Platinum Refractory Subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months | 9.76 [6.51 to 11.37] | 9.59 [7.13 to 14.26]
Statistical Analysis 1: Comparison: Treatment A - Platinum Refractory Subgroup vs Treatment B - Platinum Refractory Subgroup; Test type: Superiority; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.81 to 1.45] — computed using a cox proportional hazard model stratified by randomization PDL-1 and HPV status

10. Secondary Outcome: Overall Survival (OS) - Platinum Eligible Subgroup
Description: as for outcome 8
Time Frame: From randomization to death. Approximately 63 Months
Population: All Randomized Participants - Platinum Eligible Subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
Months | 9.71 [7.43 to 12.62] | 12.91 [9.33 to 22.01]
Statistical Analysis 1: Comparison: Treatment A - Platinum Eligible Subgroup vs Treatment B - Platinum Eligible Subgroup; Test type: Superiority; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.81 to 1.61] — computed using a cox proportional hazard model stratified by randomization PDL-1 and HPV status

11. Secondary Outcome: ORR - Platinum Eligible Subgroup Based on HPV p-16 Status
Description: ORR is defined as the best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized participants for each treatment group.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to end of study. Approximately 63 Months
Population: All Randomized Participants - Platinum Eligible Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
percentage of participants
  Positive: number analyzed (Participants) | 35 | 17
  Positive | 20.0 [8.4 to 36.9] | 41.2 [18.4 to 67.1]
  Negative: number analyzed (Participants) | 88 | 44
  Negative | 20.5 [12.6 to 30.4] | 25.0 [13.2 to 40.3]

12. Secondary Outcome: ORR - Platinum Eligible Subgroup Based on Tumor Mutation Burden (TMB) Biomarker
Description: ORR is defined as the best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized participants for each treatment group.
  Tumor Mutational Burden (TMB) refers to the number of nonsynonymous somatic mutations that exist within a tumor's genome as measured by the Foundation One CDx panel at Foundation Medicine. The analysis was done on subjects with baseline tumor mutation burden by a cutoff of 7 mutations/megabase (mut/Mb) and 10 mut/Mb
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to end of study. Approximately 63 Months
Population: All Randomized Participants - Platinum Eligible Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
percentage of participants
  TMB < 7: number analyzed (Participants) | 59 | 26
  TMB < 7 | 10.2 [3.8 to 20.8] | 30.8 [14.3 to 51.8]
  TMB ≥ 7: number analyzed (Participants) | 38 | 21
  TMB ≥ 7 | 34.2 [19.6 to 51.4] | 28.6 [11.3 to 52.2]
  TMB < 10: number analyzed (Participants) | 81 | 35
  TMB < 10 | 17.3 [9.8 to 27.3] | 28.6 [14.6 to 46.3]
  TMB ≥ 10: number analyzed (Participants) | 16 | 12
  TMB ≥ 10 | 31.3 [11.0 to 58.7] | 33.3 [9.9 to 65.1]
  TMB Not Reported: number analyzed (Participants) | 26 | 14
  TMB Not Reported | 23.1 [9.0 to 43.6] | 28.6 [8.4 to 58.1]

13. Secondary Outcome: ORR - Platinum Refractory Subgroup Based on HPV p-16 Status
Description: as for outcome 11
Time Frame: From randomization to end of study. Approximately 63 Months
Population: All Randomized Participants - Platinum Refractory Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
percentage of participants
  OROPHARYNGEAL HPV P-16 POSITIVE: number analyzed (Participants) | 30 | 16
  OROPHARYNGEAL HPV P-16 POSITIVE | 23.3 [9.9 to 42.3] | 37.5 [15.2 to 64.6]
  OROPHARYNGEAL HPV P-16 NEGATIVE/ NON-OROPHARYNGEAL: number analyzed (Participants) | 129 | 66
  OROPHARYNGEAL HPV P-16 NEGATIVE/ NON-OROPHARYNGEAL | 12.4 [7.3 to 19.4] | 16.7 [8.6 to 27.9]

14. Secondary Outcome: ORR - Platinum Refractory Subgroup Based on Tumor Mutation Burden (TMB) Biomarker
Description: as for outcome 12
Time Frame: From randomization to end of study. Approximately 63 Months
Population: All Randomized Participants - Platinum Refractory Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
percentage of participants
  TMB < 7: number analyzed (Participants) | 67 | 39
  TMB < 7 | 9.0 [3.4 to 18.5] | 20.5 [9.3 to 36.5]
  TMB ≥ 7: number analyzed (Participants) | 43 | 21
  TMB ≥ 7 | 23.3 [11.8 to 38.6] | 19.0 [5.4 to 41.9]
  TMB < 10: number analyzed (Participants) | 91 | 49
  TMB < 10 | 11.0 [5.4 to 19.3] | 22.4 [11.8 to 36.6]
  TMB ≥ 10: number analyzed (Participants) | 19 | 11
  TMB ≥ 10 | 31.6 [12.6 to 56.6] | 18.2 [2.3 to 51.8]
  TMB Not Reported: number analyzed (Participants) | 49 | 22
  TMB Not Reported | 14.3 [5.9 to 27.2] | 18.2 [5.2 to 40.3]

15. Secondary Outcome: Duration of Response (DOR) - Platinum Refractory Subgroup Based on HPV p-16 Status
Description: as for outcome 2
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: All treated participants in the Platinum Refractory subgroup with a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 21 | 15
Months
  HPV p-16 Positive: number analyzed (Participants) | 7 | 6
  HPV p-16 Positive | NA [6.87 to NA] — Insufficient number of events to calculate median and upper limit number. | 11.10 [4.17 to 14.9]
  HPV p-16 Negative: number analyzed (Participants) | 16 | 11
  HPV p-16 Negative | 39.43 [26.71 to NA] — Insufficient number of events to calculate upper limit number. | 8.34 [2.79 to NA] — Insufficient number of events to calculate upper limit number.

16. Secondary Outcome: Duration of Response (DOR) - Platinum Refractory Subgroup Based on Tumor Mutation Burden (TMB) Status
Description: The time between the date of first confirmed response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first.
  Tumor Mutational Burden (TMB) refers to the number of nonsynonymous somatic mutations that exist within a tumor's genome as measured by the Foundation One CDx panel at Foundation Medicine. The analysis was done on subjects with baseline tumor mutation burden by a cutoff of 7 mutations/megabase (mut/Mb) and 10 mut/Mb
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: All treated participants in the Platinum Refractory subgroup with a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 21 | 15
Months
  TMB: <7: number analyzed (Participants) | 6 | 8
  TMB: <7 | NA [11.01 to NA] — Insufficient number of events to calculate median and upper limit number. | 11.14 [2.69 to NA] — Insufficient number of events to calculate upper limit number.
  TMB ≥ 7: number analyzed (Participants) | 10 | 4
  TMB ≥ 7 | 38.67 [3.06 to 39.43] | 8.59 [2.79 to NA] — Insufficient number of events to calculate upper limit number.
  TMB: <10: number analyzed (Participants) | 10 | 11
  TMB: <10 | NA [3.06 to NA] — Insufficient number of events to calculate upper limit number and median | 11.14 [4.17 to NA] — Insufficient number of events to calculate upper limit number.
  TMB: ≥ 10: number analyzed (Participants) | 6 | 2
  TMB: ≥ 10 | 38.67 [6.87 to 38.67] | 7.54 [2.79 to 12.29]
  TMB: Not Reported: number analyzed (Participants) | 6 | 4
  TMB: Not Reported | 26.71 [6.93 to 26.71] | 8.21 [4.14 to 14.29]

17. Secondary Outcome: Progression Free Survival (PFS) - Platinum Refractory Subgroup Based on HPV p-16 Status
Description: as for outcome 6
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum Refractory subgroup all randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months
  Postive: number analyzed (Participants) | 30 | 16
  Postive | 4.11 [1.81 to 8.31] | 6.70 [1.28 to 13.67]
  Negative: number analyzed (Participants) | 129 | 66
  Negative | 1.84 [1.41 to 2.63] | 1.94 [1.41 to 3.02]

18. Secondary Outcome: Progression Free Survival (PFS) - Platinum Refractory Subgroup Based on Tumor Mutation Burden (TMB) Status
Description: the time from randomization to the date of first documented disease progression, or death due to any cause, whichever occurs first.
  Tumor Mutational Burden (TMB) refers to the number of nonsynonymous somatic mutations that exist within a tumor's genome as measured by the Foundation One CDx panel at Foundation Medicine. The analysis was done on subjects with baseline tumor mutation burden by a cutoff of 7 mutations/megabase (mut/Mb) and 10 mut/Mb
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum Refractory subgroup all randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months
  TMB: < 7: number analyzed (Participants) | 67 | 39
  TMB: < 7 | 1.45 [1.38 to 2.60] | 2.50 [1.41 to 5.26]
  TMB: ≥ 7: number analyzed (Participants) | 43 | 21
  TMB: ≥ 7 | 2.76 [1.45 to 4.11] | 1.54 [1.25 to 4.07]
  TMB: < 10: number analyzed (Participants) | 91 | 49
  TMB: < 10 | 1.68 [1.41 to 2.60] | 2.50 [1.41 to 4.24]
  TMB: ≥ 10: number analyzed (Participants) | 19 | 11
  TMB: ≥ 10 | 2.81 [1.38 to 9.69] | 1.41 [1.25 to 4.07]
  TMB: Not Reported: number analyzed (Participants) | 49 | 22
  TMB: Not Reported | 2.66 [1.45 to 2.92] | 2.92 [1.28 to 7.00]

19. Secondary Outcome: Overall Survival (OS) - Platinum Refractory Subgroup Based on HPV p-16 Status
Description: as for outcome 8
Time Frame: From randomization to death. Approximately 63 Months
Population: All Randomized Participants - Platinum Refractory Subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months
  Positive: number analyzed (Participants) | 30 | 16
  Positive | 13.93 [5.98 to 33.81] | 14.32 [6.28 to 44.88]
  Negative: number analyzed (Participants) | 129 | 66
  Negative | 9.36 [5.98 to 10.87] | 9.59 [6.93 to 13.40]

20. Secondary Outcome: Overall Survival (OS) - Platinum Refractory Subgroup Based on Tumor Mutation Burden (TMB) Status
Description: Overall survival was defined as the time from randomization to the date of death from any cause. Participants were censored at the date they were last known to be alive and at the date of randomization if they were randomized but had no follow-up.
  Tumor Mutational Burden (TMB) refers to the number of nonsynonymous somatic mutations that exist within a tumor's genome as measured by the Foundation One CDx panel at Foundation Medicine. The analysis was done on subjects with baseline tumor mutation burden by a cutoff of 7 mutations/megabase (mut/Mb) and 10 mut/Mb
Time Frame: From randomization to death. Approximately 63 Months
Population: All Randomized Participants - Platinum Refractory Subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months
  TMB: <7: number analyzed (Participants) | 67 | 39
  TMB: <7 | 5.78 [3.45 to 9.76] | 8.77 [4.14 to 16.66]
  TMB: ≥ 7: number analyzed (Participants) | 43 | 21
  TMB: ≥ 7 | 11.37 [6.41 to 16.95] | 7.16 [6.28 to 12.29]
  TMB: < 10: number analyzed (Participants) | 91 | 49
  TMB: < 10 | 7.52 [4.96 to 11.27] | 8.31 [4.90 to 13.04]
  TMB: ≥10: number analyzed (Participants) | 19 | 11
  TMB: ≥10 | 6.51 [2.50 to 41.33] | 9.26 [1.35 to 17.51]
  Not Reported: number analyzed (Participants) | 49 | 22
  Not Reported | 13.86 [9.53 to 17318] | 20.01 [7.56 to 23.46]

21. Secondary Outcome: Overall Survival (OS) - Platinum Eligible Subgroup Based on HPV p-16 Status
Description: as for outcome 8
Time Frame: From randomization to death. Approximately 63 Months
Population: All Randomized Participants - Platinum Eligible Subgroup
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Treatment B - Platinum Eligible Subgroup: Participants with histologically confirmed Squamous Cell Carcinoma of the Head and Neck (SCCHN) who are platinum naive or have recurred 6 months or more after completion of previous platinum-based chemotherapy.
  Treated with Nivolumab 3 mg/kg Q2W + Ipilimumab 1 mg/kg Q6W
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
Months
  Positive: number analyzed (Participants) | 35 | 17
  Positive | 16.66 [8.54 to 28.06] | 33.74 [12.91 to NA] — Insufficient number of events to calculate upper limit number.
  Negative: number analyzed (Participants) | 88 | 44
  Negative | 7.79 [5.06 to 12.39] | 9.46 [5.32 to 14.00]

22. Secondary Outcome: Overall Survival (OS) - Platinum Eligible Subgroup Based on Tumor Mutation Burden (TMB) Status
Description: as for outcome 20
Time Frame: From randomization to death. Approximately 63 Months
Population: All Randomized Participants - Platinum Eligible Subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
Months
  TMB: <7: number analyzed (Participants) | 59 | 26
  TMB: <7 | 7.56 [4.83 to 12.25] | 18.27 [4.04 to 33.74]
  TMB: ≥ 7: number analyzed (Participants) | 38 | 21
  TMB: ≥ 7 | 16.30 [9.43 to 36.30] | 13.08 [8.28 to 38.11]
  TMB: < 10: number analyzed (Participants) | 81 | 35
  TMB: < 10 | 9.99 [6.41 to 12.62] | 15.01 [7.62 to 27.47]
  TMB: ≥10: number analyzed (Participants) | 16 | 12
  TMB: ≥10 | 16.72 [4.47 to NA] — upper limit not calculable | 14.77 [2.83 to NA] — upper limit not calculable
  Not Reported: number analyzed (Participants) | 26 | 14
  Not Reported | 8.00 [3.84 to 26.12] | 9.71 [2.56 to 18.79]

23. Secondary Outcome: Progression Free Survival (PFS) - Platinum Eligible Subgroup Based on Tumor Mutation Burden (TMB) Status
Description: as for outcome 18
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum eligible subgroup all randomized
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
Months
  TMB: < 7: number analyzed (Participants) | 59 | 26
  TMB: < 7 | 2.63 [1.45 to 3.06] | 2.92 [1.38 to 9.59]
  TMB: ≥ 7: number analyzed (Participants) | 38 | 21
  TMB: ≥ 7 | 5.82 [1.45 to 12.42] | 2.83 [1.41 to 13.01]
  TMB: < 10: number analyzed (Participants) | 81 | 35
  TMB: < 10 | 2.63 [1.45 to 3.06] | 2.99 [1.41 to 13.01]
  TMB: ≥ 10: number analyzed (Participants) | 16 | 12
  TMB: ≥ 10 | 6.97 [1.41 to NA] — Insufficient number of events to calculate upper limit number. | 2.76 [0.72 to 27.60]
  TMB: Not Reported: number analyzed (Participants) | 26 | 14
  TMB: Not Reported | 2.71 [1.45 to 8.48] | 3.10 [1.38 to 9.82]

24. Secondary Outcome: Progression Free Survival (PFS) - Platinum Eligible Subgroup Based on HPV p-16 Status
Description: as for outcome 6
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum eligible subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
Months
  Postive: number analyzed (Participants) | 35 | 17
  Postive | 2.92 [1.41 to 6.60] | 6.83 [1.38 to 49.84]
  Negative: number analyzed (Participants) | 88 | 44
  Negative | 2.66 [1.51 to 4.14] | 2.83 [1.51 to 4.24]

25. Secondary Outcome: Duration of Response (DOR) - Platinum Eligible Subgroup Based on HPV p-16 Status
Description: The time between the date of first confirmed response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: All treated participants in the Platinum Eligible subgroup with a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 25 | 18
Months
  Positive: number analyzed (Participants) | 7 | 7
  Positive | 33.84 [4.14 to NA] — Insufficient number of events to calculate upper limit number. | 48.49 [5.49 to NA] — Insufficient number of events to calculate upper limit number.
  Negative: number analyzed (Participants) | 18 | 11
  Negative | 27.04 [10.97 to NA] — Insufficient number of events to calculate upper limit number. | 19.32 [4.11 to NA] — Insufficient number of events to calculate upper limit number.

26. Secondary Outcome: Duration of Response (DOR) - Platinum Eligible Subgroup Based on Tumor Mutation Burden (TMB) Status
Description: The time between the date of first confirmed response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first.
  Tumor Mutational Burden (TMB) refers to the number of nonsynonymous somatic mutations that exist within a tumor's genome as measured by the Foundation One CDx panel at Foundation Medicine. The analysis was done on subjects with baseline tumor mutation burden by a cutoff of 7 mutations/megabase (mut/Mb) and 10 mut/Mb.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: All treated participants in the Platinum eligible subgroup with a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 25 | 18
Months
  TMB: <7: number analyzed (Participants) | 6 | 8
  TMB: <7 | 10.97 [4.14 to 35.55] | NA [5.52 to NA] — Insufficient number of events to calculate upper limit number and median
  TMB ≥ 7: number analyzed (Participants) | 13 | 6
  TMB ≥ 7 | 24.11 [10.97 to NA] — Insufficient number of events to calculate upper limit number. | 19.32 [5.49 to 24.61]
  TMB: <10: number analyzed (Participants) | 14 | 10
  TMB: <10 | 13.67 [8.28 to 35.55] | NA [5.52 to NA] — Insufficient number of events to calculate upper limit number and median
  TMB: ≥ 10: number analyzed (Participants) | 5 | 4
  TMB: ≥ 10 | NA [5.78 to NA] — Insufficient number of events to calculate upper limit number and median | 19.32 [5.49 to 24.61]
  TMB: Not Reported: number analyzed (Participants) | 6 | 4
  TMB: Not Reported | NA [27.04 to NA] — Insufficient number of events to calculate upper limit number and median. | 48.49 [4.11 to NA] — Insufficient number of events to calculate upper limit number.

27. Secondary Outcome: Duration of Response (DOR) - Platinum Refractory Subgroup Based on PD-L1 Status
Description: The time between the date of first confirmed response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first.
  Tumor PD-L1 expression was defined as the percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 IHC assay.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: All treated participants in the Platinum refractory subgroup with a response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 21 | 15
Months
  PD-L1: ≥ 1%: number analyzed (Participants) | 18 | 9
  PD-L1: ≥ 1% | 39.43 [11.01 to NA] — Insufficient number of events to calculate upper limit number. | 8.34 [2.79 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: < 25%: number analyzed (Participants) | 13 | 12
  PD-L1: < 25% | 39.43 [6.87 to NA] — Insufficient number of events to calculate upper limit number. | 11.10 [4.17 to 38.51]
  PD-L1: ≥ 25%: number analyzed (Participants) | 9 | 5
  PD-L1: ≥ 25% | NA [6.93 to NA] — Insufficient number of events to calculate upper limit number and median | 8.34 [2.79 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: <50%: number analyzed (Participants) | 17 | 15
  PD-L1: <50% | NA [26.71 to NA] — Insufficient number of events to calculate upper limit number and median | 11.14 [4.17 to 38.51]
  PD-L1: > 50%: number analyzed (Participants) | 5 | 2
  PD-L1: > 50% | NA [6.93 to NA] — Insufficient number of events to calculate upper limit number and median | 6.24 [4.14 to 8.34]
  PD-L1: 1 - < 25%: number analyzed (Participants) | 9 | 4
  PD-L1: 1 - < 25% | 39.43 [3.06 to 39.43] | NA [4.17 to NA] — Insufficient number of events to calculate upper limit number and median
  PD-L1: Unquantifiable: number analyzed (Participants) | 1 | 0
  PD-L1: Unquantifiable | 38.67 [NA to NA] — Insufficient number of events to calculate upper limit number and lower limit number |

28. Secondary Outcome: ORR - Platinum Refractory Subgroup Based on PD-L1 Expression
Description: ORR is defined as the best overall response (BOR) of a complete response (CR) or partial response (PR) divided by the number of randomized participants for each treatment group.
  Tumor PD-L1 expression was defined as the percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 IHC assay
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes(whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From randomization to end of study. Approximately 63 Months
Population: Platinum Refractory subgroup
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Percentage of Participants
  <1%: number analyzed (Participants) | 52 | 31
  <1% | 7.7 [2.1 to 18.5] | 25.8 [11.9 to 44.6]
  PD-L1: ≥ 1%: number analyzed (Participants) | 92 | 46
  PD-L1: ≥ 1% | 19.6 [12.0 to 29.1] | 19.6 [9.4 to 33.9]
  PD-L1: < 25%: number analyzed (Participants) | 117 | 57
  PD-L1: < 25% | 11.1 [6.1 to 18.3] | 21.1 [11.4 to 33.9]
  PD-L1: ≥ 25%: number analyzed (Participants) | 27 | 20
  PD-L1: ≥ 25% | 33.3 [16.5 to 54.0] | 25.0 [8.7 to 49.1]
  PD-L1: <50%: number analyzed (Participants) | 129 | 66
  PD-L1: <50% | 13.2 [7.9 to 20.3] | 22.7 [13.3 to 34.7]
  PD-L1: > 50%: number analyzed (Participants) | 15 | 11
  PD-L1: > 50% | 33.3 [11.8 to 61.6] | 18.2 [2.3 to 51.8]
  PD-L1: 1 - < 25%: number analyzed (Participants) | 65 | 26
  PD-L1: 1 - < 25% | 13.8 [6.5 to 24.7] | 15.4 [4.4 to 34.9]
  without quantifiable PD-L1 expression at baseline: number analyzed (Participants) | 15 | 5
  without quantifiable PD-L1 expression at baseline | NA [NA to NA] — Not reported when sample size is less than 10 subjects for the subgroup category | NA [NA to NA] — Not reported when sample size is less than 10 subjects for the subgroup category

29. Secondary Outcome: Overall Survival (OS) - Platinum Refractory Subgroup Based on PD-L1 Status
Description: Overall survival was defined as the time from randomization to the date of death from any cause. Participants were censored at the date they were last known to be alive and at the date of randomization if they were randomized but had no follow-up.
  Tumor PD-L1 expression was defined as the percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 IHC assay
Time Frame: From randomization to death. Approximately 63 Months
Population: Platinum refractory subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months
  <1%: number analyzed (Participants) | 52 | 31
  <1% | 9.53 [6.31 to 12.62] | 12.29 [6.08 to 20.27]
  PD-L1: ≥ 1%: number analyzed (Participants) | 92 | 46
  PD-L1: ≥ 1% | 10.22 [5.95 to 14.52] | 9.02 [6.74 to 13.34]
  PD-L1: < 25%: number analyzed (Participants) | 117 | 57
  PD-L1: < 25% | 9.95 [7.26 to 11.37] | 8.77 [6.28 to 14.78]
  PD-L1: ≥ 25%: number analyzed (Participants) | 27 | 20
  PD-L1: ≥ 25% | 5.78 [2.43 to 48.69] | 10.23 [7.03 to 16.66]
  PD-L1: <50%: number analyzed (Participants) | 129 | 66
  PD-L1: <50% | 9.76 [6.51 to 11.37] | 10.61 [6.74 to 14.26]
  PD-L1: > 50%: number analyzed (Participants) | 15 | 11
  PD-L1: > 50% | 26.02 [2.43 to 48.69] | 7.33 [1.51 to 16.66]
  PD-L1: 1 - < 25%: number analyzed (Participants) | 65 | 26
  PD-L1: 1 - < 25% | 10.32 [5.98 to 14.32] | 7.56 [4.86 to 17.51]
  Without quantifiable PD-L1 expression at baseline: number analyzed (Participants) | 15 | 5
  Without quantifiable PD-L1 expression at baseline | 6.93 [1.71 to 14.16] | 28.09 [7.56 to 44.88]

30. Secondary Outcome: Progression Free Survival (PFS) - Platinum Refractory Subgroup Based on PD-L1 Status
Description: The time from randomization to the date of first documented disease progression, or death due to any cause, whichever occurs first.
  Tumor PD-L1 expression was defined as the percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 IHC assay.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum Refractory subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
Months
  <1%: number analyzed (Participants) | 52 | 31
  <1% | 2.60 [1.41 to 2.86] | 2.96 [1.38 to 5.32]
  PD-L1: ≥ 1%: number analyzed (Participants) | 92 | 46
  PD-L1: ≥ 1% | 2.60 [1.45 to 2.83] | 2.60 [1.41 to 4.11]
  PD-L1: < 25%: number analyzed (Participants) | 117 | 57
  PD-L1: < 25% | 2.60 [1.45 to 2.83] | 2.79 [1.41 to 4.01]
  PD-L1: ≥ 25%: number analyzed (Participants) | 27 | 20
  PD-L1: ≥ 25% | 2.12 [1.38 to 13.77] | 1.54 [1.25 to 7.03]
  PD-L1: <50%: number analyzed (Participants) | 129 | 66
  PD-L1: <50% | 2.60 [1.45 to 2.79] | 2.79 [1.54 to 4.07]
  PD-L1: > 50%: number analyzed (Participants) | 15 | 11
  PD-L1: > 50% | 2.79 [0.59 to 13.77] | 1.54 [0.66 to 7.03]
  PD-L1: 1 - < 25%: number analyzed (Participants) | 65 | 26
  PD-L1: 1 - < 25% | 2.66 [1.45 to 2.83] | 2.60 [1.38 to 4.07]
  Without Quantifiable PD-L1 expression at Baseline: number analyzed (Participants) | 15 | 5
  Without Quantifiable PD-L1 expression at Baseline | 2.17 [1.08 to 2.66] | 1.71 [1.22 to NA] — insufficient number of participants with an event to calculate

31. Secondary Outcome: Duration of Response (DOR) - Platinum Eligible Subgroup Based on PD-L1 Status
Description: The time between the date of first confirmed response to the date of the first documented tumor progression, or death due to any cause, whichever occurs first.
  Tumor PD-L1 expression was defined as the percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 IHC assay
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum Eligible Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 25 | 18
Months
  PD-L1: ≥ 1%: number analyzed (Participants) | 14 | 10
  PD-L1: ≥ 1% | 33.84 [8.28 to NA] — Insufficient number of events to calculate upper limit number. | 24.61 [4.11 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: < 25%: number analyzed (Participants) | 13 | 9
  PD-L1: < 25% | 13.17 [4.17 to 35.55] | 12.42 [4.11 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: ≥ 25%: number analyzed (Participants) | 9 | 6
  PD-L1: ≥ 25% | NA [8.28 to NA] — Insufficient number of events to calculate upper limit number and median | NA [24.61 to NA] — Insufficient number of events to calculate upper limit number and median
  PD-L1: <50%: number analyzed (Participants) | 16 | 10
  PD-L1: <50% | 13.67 [5.78 to 35.55] | 15.87 [4.11 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: > 50%: number analyzed (Participants) | 6 | 5
  PD-L1: > 50% | NA [33.84 to NA] — Insufficient number of events to calculate upper limit number and median | NA [24.61 to NA] — Insufficient number of events to calculate upper limit number and median
  PD-L1: 1 - < 25%: number analyzed (Participants) | 5 | 4
  PD-L1: 1 - < 25% | 13.13 [4.14 to NA] — Insufficient number of events to calculate upper limit number. | 6.21 [4.11 to 12.42]
  PD-L1: Unquantifiable: number analyzed (Participants) | 3 | 3
  PD-L1: Unquantifiable | NA [27.04 to NA] — Insufficient number of events to calculate upper limit number and median | 28.99 [9.49 to 48.49]

32. Secondary Outcome: ORR - Platinum Eligible Subgroup Based on PD-L1 Expression
Description: as for outcome 28
Time Frame: From randomization to end of study. Approximately 63 Months
Population: Platinum Eligible Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
percentage of participants
  <1%: number analyzed (Participants) | 51 | 23
  <1% | 15.7 [7.0 to 28.6] | 21.7 [7.5 to 43.7]
  PD-L1: ≥ 1%: number analyzed (Participants) | 65 | 33
  PD-L1: ≥ 1% | 21.5 [12.3 to 33.5] | 30.3 [15.6 to 48.7]
  PD-L1: < 25%: number analyzed (Participants) | 87 | 37
  PD-L1: < 25% | 14.9 [8.2 to 24.2] | 24.3 [11.8 to 41.2]
  PD-L1: ≥ 25%: number analyzed (Participants) | 29 | 19
  PD-L1: ≥ 25% | 31.0 [15.3 to 50.8] | 31.6 [12.6 to 56.6]
  PD-L1: <50%: number analyzed (Participants) | 96 | 41
  PD-L1: <50% | 16.7 [9.8 to 25.6] | 24.4 [12.4 to 40.3]
  PD-L1: > 50%: number analyzed (Participants) | 20 | 15
  PD-L1: > 50% | 30.0 [11.9 to 54.3] | 33.3 [11.8 to 61.6]
  PD-L1: 1 - < 25%: number analyzed (Participants) | 36 | 14
  PD-L1: 1 - < 25% | 13.9 [4.7 to 29.5] | 28.6 [8.4 to 58.1]
  Without quantifiable PD-L1 expression at baseline: number analyzed (Participants) | 7 | 5
  Without quantifiable PD-L1 expression at baseline | NA [NA to NA] — Not reported when sample size is less than 10 subjects for the subgroup category,CI not calculable | NA [NA to NA] — Not reported when sample size is less than 10 subjects for the subgroup category, CI not calculable

33. Secondary Outcome: Overall Survival (OS) - Platinum Eligible Subgroup Based on PD-L1 Status
Description: as for outcome 29
Time Frame: From randomization to death. Approximately 63 Months
Population: Platinum Eligible Subgroup
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
months
  <1%: number analyzed (Participants) | 51 | 23
  <1% | 12.52 [8.21 to 17.68] | 11.17 [3.42 to 21.52]
  PD-L1: ≥ 1%: number analyzed (Participants) | 65 | 33
  PD-L1: ≥ 1% | 7.56 [5.06 to 11.24] | 14.00 [7.62 to 23.66]
  PD-L1: < 25%: number analyzed (Participants) | 87 | 37
  PD-L1: < 25% | 8.72 [5.91 to 12.25] | 11.17 [5.32 to 21.52]
  PD-L1: ≥ 25%: number analyzed (Participants) | 29 | 19
  PD-L1: ≥ 25% | 12.39 [5.06 to 36.30] | 14.00 [6.34 to 38.74]
  PD-L1: <50%: number analyzed (Participants) | 96 | 41
  PD-L1: <50% | 9.10 [6.57 to 12.62] | 9.92 [4.04 to 18.79]
  PD-L1: > 50%: number analyzed (Participants) | 20 | 15
  PD-L1: > 50% | 9.40 [4.11 to 36.30] | 15.01 [7.62 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: 1 - < 25%: number analyzed (Participants) | 36 | 14
  PD-L1: 1 - < 25% | 6.16 [4.57 to 8.11] | 8.48 [2.83 to 22.41]
  Without quantifiable PD-L1 expression at baseline: number analyzed (Participants) | 7 | 5
  Without quantifiable PD-L1 expression at baseline | 26.12 [1.64 to NA] — Insufficient number of events to calculate upper limit number. | 33.74 [5.72 to NA] — Insufficient number of events to calculate upper limit number.

34. Secondary Outcome: Progression Free Survival (PFS) - Platinum Eligible Subgroup Based on PD-L1 Status
Description: The time from randomization to the date of first documented disease progression, or death due to any cause, whichever occurs first.
  Tumor PD-L1 expression was defined as the percent of tumor cell membrane staining in a minimum of 100 evaluable tumor cells per validated Dako PD-L1 IHC assay
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum eligible subgroup
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
Number analyzed (Participants) | 123 | 61
Months
  <1%: number analyzed (Participants) | 51 | 23
  <1% | 2.61 [1.38 to 5.78] | 2.73 [1.41 to 9.82]
  PD-L1: ≥ 1%: number analyzed (Participants) | 65 | 33
  PD-L1: ≥ 1% | 2.89 [1.51 to 4.21] | 2.99 [1.38 to 5.65]
  PD-L1: < 25%: number analyzed (Participants) | 87 | 37
  PD-L1: < 25% | 2.37 [1.41 to 2.76] | 2.76 [1.41 to 5.65]
  PD-L1: ≥ 25%: number analyzed (Participants) | 29 | 19
  PD-L1: ≥ 25% | 5.75 [3.71 to 16.59] | 2.99 [1.38 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: <50%: number analyzed (Participants) | 96 | 41
  PD-L1: <50% | 2.55 [1.45 to 2.89] | 2.76 [1.41 to 5.65]
  PD-L1: > 50%: number analyzed (Participants) | 20 | 15
  PD-L1: > 50% | 4.21 [2.79 to NA] — Insufficient number of events to calculate upper limit number. | 2.99 [1.38 to NA] — Insufficient number of events to calculate upper limit number.
  PD-L1: 1 - < 25%: number analyzed (Participants) | 36 | 14
  PD-L1: 1 - < 25% | 1.51 [1.41 to 2.86] | 3.10 [1.28 to 8.28]
  Without quantifiable PD-L1 expression at baseline: number analyzed (Participants) | 7 | 5
  Without quantifiable PD-L1 expression at baseline | 6.47 [1.51 to NA] — Insufficient number of events to calculate upper limit number. | 13.73 [1.28 to 49.84]

35. Post Hoc Outcome: Objective Response Rate (ORR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Refractory Subgroup - Post Hoc Analysis
Description: as for outcome 1
Time Frame: From randomization to end of study. Approximately 63 Months
Population: All Randomized Participants - Platinum Refractory Subgroup
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 159 | 82
percentage of participants | 14.5 [9.4 to 20.9] | 20.7 [12.6 to 31.1]
Statistical Analysis 1: Comparison: Treatment A - Platinum Refractory Subgroup vs Treatment B - Platinum Refractory Subgroup; Treatment A over Treatment B; Test type: Superiority; Mantel Haenszel; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.32 to 1.29]

36. Post Hoc Outcome: Duration of Response (DOR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Refractory Subgroup - Post Hoc Analysis
Description: as for outcome 25
Time Frame: From randomization to disease progression or death. Approximately 63 Months
Population: Platinum Refractory Responders
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 23 | 17
Months | 39.43 [26.71 to NA] — Upper Limit not calculable | 11.07 [4.17 to 38.51]

37. Post Hoc Outcome: Time to Response (TTR) as Determined by Blinded Independent Central Review (BIRC) - Platinum Refractory Subgroup - Post Hoc Analysis
Description: as for outcome 3
Time Frame: From randomization to a confirmed response. Approximately 35 Months
Population: Platinum refractory responders
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup
Number analyzed (Participants) | 23 | 17
Months | 2.63 [1.1 to 34.3] | 1.71 [1.2 to 7.7]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately 32 months All-Cause mortality (From randomization to end of study): Approximately 63 months
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Treatment A - Platinum Refractory Subgroup | Treatment B - Platinum Refractory Subgroup | Treatment A - Platinum Eligible Subgroup | Treatment B - Platinum Eligible Subgroup
All-Cause Mortality (participants affected / at risk) | 131/159 | 71/82 | 102/123 | 49/61
Serious Adverse Events (participants affected / at risk) | 103/158 | 52/82 | 89/122 | 35/61
Other Adverse Events (participants affected / at risk) | 139/158 | 76/82 | 118/122 | 54/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A - Platinum Refractory Subgroup (N=158) | Treatment B - Platinum Refractory Subgroup (N=82) | Treatment A - Platinum Eligible Subgroup (N=122) | Treatment B - Platinum Eligible Subgroup (N=61)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 2 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 0 | 0 | 0 | 1
Hypophysitis (Endocrine disorders) | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Autoimmune colitis (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 4 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 0 | 5 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 3 | 1 | 2 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 2 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Oesophageal fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 3 | 2 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 0 | 0 | 1
Drug intolerance (General disorders) | 1 | 0 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 3 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0
Impaired healing (General disorders) | 0 | 0 | 1 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0 | 2 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 1 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 3 | 0
Swelling (General disorders) | 1 | 0 | 0 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0 | 0
Empyema (Infections and infestations) | 0 | 0 | 0 | 1
Encephalitis (Infections and infestations) | 0 | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Epiglottitis (Infections and infestations) | 0 | 0 | 1 | 0
Focal peritonitis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Hepatic infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0
Infective myositis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Ludwig angina (Infections and infestations) | 0 | 0 | 1 | 0
Lymph node abscess (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Oral infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 18 | 5 | 10 | 4
Pneumonia aspiration (Infections and infestations) | 2 | 0 | 3 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 2 | 0 | 0
Staphylococcal scalded skin syndrome (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Tracheitis (Infections and infestations) | 2 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Tracheostomy infection (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2 | 1
Vascular access site infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral myocarditis (Infections and infestations) | 0 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Vasoplegia syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 6 | 2 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 61 | 25 | 47 | 16
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Carotid aneurysm rupture (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 2
Device leakage (Product Issues) | 2 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 2 | 0
Autoimmune lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 4 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 1 | 2 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral venous disease (Vascular disorders) | 0 | 0 | 2 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A - Platinum Refractory Subgroup (N=158) | Treatment B - Platinum Refractory Subgroup (N=82) | Treatment A - Platinum Eligible Subgroup (N=122) | Treatment B - Platinum Eligible Subgroup (N=61)
Anaemia (Blood and lymphatic system disorders) | 41 | 33 | 30 | 15
Lymphopenia (Blood and lymphatic system disorders) | 12 | 3 | 0 | 2
Hyperthyroidism (Endocrine disorders) | 12 | 4 | 11 | 1
Hypothyroidism (Endocrine disorders) | 28 | 10 | 23 | 12
Abdominal pain (Gastrointestinal disorders) | 8 | 5 | 10 | 4
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 4 | 5
Constipation (Gastrointestinal disorders) | 24 | 14 | 26 | 9
Diarrhoea (Gastrointestinal disorders) | 33 | 17 | 27 | 15
Dry mouth (Gastrointestinal disorders) | 11 | 4 | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 0 | 7 | 3
Dysphagia (Gastrointestinal disorders) | 16 | 10 | 18 | 7
Nausea (Gastrointestinal disorders) | 31 | 18 | 28 | 13
Stomatitis (Gastrointestinal disorders) | 2 | 5 | 6 | 1
Vomiting (Gastrointestinal disorders) | 18 | 9 | 14 | 5
Asthenia (General disorders) | 27 | 14 | 13 | 7
Chills (General disorders) | 2 | 0 | 7 | 0
Face oedema (General disorders) | 9 | 3 | 7 | 2
Fatigue (General disorders) | 29 | 21 | 46 | 22
Mucosal inflammation (General disorders) | 9 | 4 | 8 | 2
Oedema peripheral (General disorders) | 7 | 6 | 10 | 1
Pyrexia (General disorders) | 15 | 9 | 15 | 5
Nasopharyngitis (Infections and infestations) | 2 | 1 | 6 | 4
Oral candidiasis (Infections and infestations) | 9 | 2 | 1 | 2
Pneumonia (Infections and infestations) | 10 | 5 | 8 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 4
Alanine aminotransferase increased (Investigations) | 8 | 4 | 7 | 6
Amylase increased (Investigations) | 4 | 5 | 10 | 3
Aspartate aminotransferase increased (Investigations) | 9 | 4 | 11 | 5
Blood alkaline phosphatase increased (Investigations) | 7 | 9 | 9 | 3
Blood creatinine increased (Investigations) | 11 | 10 | 7 | 5
Blood thyroid stimulating hormone increased (Investigations) | 4 | 1 | 5 | 4
Lipase increased (Investigations) | 13 | 4 | 11 | 5
Weight decreased (Investigations) | 20 | 9 | 25 | 5
Decreased appetite (Metabolism and nutrition disorders) | 21 | 17 | 25 | 8
Hypercalcaemia (Metabolism and nutrition disorders) | 18 | 10 | 11 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 4 | 5 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 7 | 8 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 2 | 12 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 6 | 9 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 11 | 14 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 9 | 18 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11 | 12 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3 | 8 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 18 | 11 | 7 | 9
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 2 | 4
Dizziness (Nervous system disorders) | 8 | 2 | 5 | 4
Headache (Nervous system disorders) | 14 | 5 | 11 | 6
Anxiety (Psychiatric disorders) | 9 | 4 | 2 | 4
Insomnia (Psychiatric disorders) | 13 | 7 | 5 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 8 | 20 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 11 | 20 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 6 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 10 | 5 | 6 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 3 | 8 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 6 | 24 | 10
Rash (Skin and subcutaneous tissue disorders) | 32 | 9 | 19 | 6
Hypertension (Vascular disorders) | 2 | 3 | 5 | 4
Hypotension (Vascular disorders) | 6 | 2 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/74/NCT02823574/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT02823574/SAP_001.pdf